CLINICAL TRIAL: NCT00642369
Title: Study of Evaluating Quetiapine in Improving Sleep Quality of Schizophrenia
Brief Title: A 4-week, Randomized, Rater-blinded, Parallel Study to Evaluate Quetiapine in Improving Sleep Quality of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang Dong Provincial Mental Health Institute (Other)
Responsible Party: Principal Investigator, Bin Zhang, sleep centre, Guang Dong Provincial Mental Health Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1443L00053
Record Dates: First submitted 2008-03-18; First posted 2008-03-25 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Polysomnograph
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Haloperidol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- quetiapine fumarate (Experimental): quetiapine fumarate was administered 25mg on the 1st day,738±41mg/day on the 14th day, and 738±48mg/day on the 28th day.
  Interventions: Drug: quetiapine fumarate
- haloperidol (Active Comparator): haloperidol was administered 2mg on the 1st day,16±7mg/day on the 14th day, and 18±6mg/day on the 28th day.
  Interventions: Drug: haloperidol

INTERVENTIONS:
Drug: quetiapine fumarate — 600-750mg/day
  Other Names: seroquel
  Arms: quetiapine fumarate
Drug: haloperidol — 6-40mg/day
  Arms: haloperidol

SUMMARY:
This study will apply polysomnography (PSG) to evaluate the effect of quetiapine fumarate on sleep architecture. Most of previous studies evaluated sleep by self-reported questionnaires during the antipsychotic treatment (clozapine, risperidone, olanzapine, et al), while only a few studies with PSG evaluation had some limitation, such as: small sample size, respective or cross-sectional, potential sleep disorders, et al. In this study, we will investigate both subjective and objective effect of quetiapine fumarate in improving sleep quality in schizophrenic patients by PSG as well as psychiatric scales. The control drug in this study is the typical antipsychotic - haloperidol. It could increase sleep duration and efficiency by mostly increasing the S2 without effect on rapid eye movement (REM) sleep and slow wave sleep (SWS). The patients will be randomised into two groups as a parallel design. This study is designed as rater blinded to reduce the bias in evaluation. It is suggested that the sedative effect of quetiapine fumarate could diminish in 2 weeks, therefore, we use 4 weeks to ensure the change of sleep quality in this study, which could be helpful for the evaluation of relative short and middle term effect of quetiapine fumarate on sleep quality.

DETAILED DESCRIPTION:
1. The objective sleep structures of quetiapine fumarate and haloperidol being used as mono-therapy respectively in the treatment of patients with acute schizophrenia are measured by the change of composite variables for PSG test (sleep stages, time in bed, total sleep time, sleep efficiency, sleep latency) from baseline to Week 4 (LOCF).
2. The subjective sleep qualities of quetiapine fumarate and haloperidol being used as mono-therapy respectively in the treatment of patients with acute schizophrenia are measured by the change of Pittsburgh Sleep Quality Inventory (PSQI) and Epworth Sleepiness Scale(ESS) from baseline to Week 4 (LOCF).
3. The clinical efficacy of quetiapine fumarate and haloperidol being used as mono-therapy respectively in the treatment of patients with acute schizophrenia are measured by the change of Positive and Negative Syndrome Scale (PANSS) and Clinical Globe Impression (CGI),and Calgary Depression Scale for Schizophrenia (CDSS) from baseline to Week 4 (LOCF).
4. The clinical safety and tolerance quetiapine fumarate and haloperidol being used as mono-therapy respectively in the treatment of patients with acute schizophrenia are measured by Treatment Emergent Symptom Scale (TESS) in day 14 and day 28.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfill all of the following criteria:

1. Provision of written informed consent by patient or his/her legal guardian
2. Hospitalized for a diagnosis of Schizophrenia paranoid subtype by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
3. Positive and Negative Syndrome Scale (PANSS) total score≥60
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chronic gonadotropin (HCG) test at enrolment
5. Able to understand and comply with the requirements of the study

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate or/and haloperidol, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
12. Organic changes was founded by brain CT
13. Involvement in the planning and conduct of the study
14. Previous enrolment or randomisation of treatment in the present study.
15. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
16. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria: unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%; admitted to hospital for treatment of DM or DM related illness in past 12 weeks; not under physician care for DM Physician responsible for patient's DM care has not indicated that patient's DM is controlled; Physician responsible for patient's DM care has not approved patient's participation in the study; has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation; for thiazolidinediones (glitazones) this period should not be less than 8 Weeks; taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks. Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
17. An absolute neutrophil count (ANC) of 1.5 x 109/L
18. Sleep disorder such as Apnea Hypopneas Syndrome, periodic leg movement syndrome and narcolepsy
19. The work time is rotate and/or often flies across the time zone
20. Use of clozapine within 28 days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Bin, Ph. D, Principal Investigator — Guang Dong Provincial Mental Health Institute
Locations (1):
- Guangdong Provincial Mental Health Institute, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine Fumarate: slow wave sleep% and rapid eye movement sleepin quetiapine fumarate treatment group
- Haloperidol: slow wave sleep% in haloperidol treatment group
Period: Overall Study
Arm/Group | Quetiapine Fumarate | Haloperidol
Started | 30 | 30
Completed | 25 | 24
Not Completed | 5 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — misdiagnosis | 0 | 1
Not completed — Lack of Efficacy | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Quetiapine Fumarate: quetiapine fumarate treatment (200-750mg/day) in 28 days
- Haloperidol: haloperidol treatment (6-40mg/day) in 28 days
- Total: Total of all reporting groups
Arm/Group | Quetiapine Fumarate | Haloperidol | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (10.1) | 27.9 (6.7) | 26.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Slow Wave Sleep
Description: The primary variable is the change of percentage of slow wave sleep (SWS) from baseline to the 28th day (LOCF).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage of slow wave sleep
Groups:
- Quetiapine Fumarate: percentage of slow wave sleep in quetiapine fumarate group
- Haloperidol: percentage of slow wave sleep in haloperidol group
Arm/Group | Quetiapine Fumarate | Haloperidol
Number analyzed (Participants) | 30 | 30
percentage of slow wave sleep
  percentage at baseline | 10.5 (5.5) | 8.6 (7.6)
  percentage on the 28th day | 9.2 (8.0) | 6.3 (5.4)
  percentage change from baseline to the 28th day | -1.4 (1.1) | -2.3 (1.8)

2. Primary Outcome: Percentage of Rapid Eye Movement Sleep
Description: The primary variable is the change of the percentage of rapid eye movement (REM)sleep from baseline to the 28th day (LOCF).
Time Frame: 28 days
Population: For the need of the statistical analysis, the study group and the control group are 30 evaluable patients respectively. Finally, in consideration of 25% un-evaluable patients after randomisation, there should be 80 patients randomised in this study with 40 patients per arm.
Measure: Mean (Standard Deviation); unit: percentage of rapid eye movement sleep
Groups:
- Quetiapine Fumarate: percentage of rapid eye movement sleep in quetiapine fumarate group
- Haloperidol: percentage of rapid eye movement sleep in haloperidol group
Arm/Group | Quetiapine Fumarate | Haloperidol
Number analyzed (Participants) | 30 | 30
percentage of rapid eye movement sleep
  percentage at baseline | 12.6 (9.1) | 13.2 (5.3)
  percentage on the 28th day | 16.4 (9.2) | 10.4 (11.3)
  percentage change from baseline to the 28th day | 3.9 (3.2) | -2.7 (2.5)

ADVERSE EVENTS:
Time Frame: 28 days.
Arm/Group | Quetiapine Fumarate | Haloperidol
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
the present study lasted for only 4 weeks. it might be too short to investigate the effect of quetiapine fumarate and haloperidol on sleep and clinical parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No